CLINICAL TRIAL: NCT02496975
Title: Oxidative Damage and Calcium-Activated Proteolytic Biomarkers After Traumatic Brain Injury and Effects of Acute Cyclosporine A
Brief Title: Traumatic Brain Injury and Effects of Acute Cyclosporine A
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Recent studies suggest that cyclosporine A has a very sharp biphasic dose-response problem that is going to make further clinical translation difficult.
Sponsor: Edward Hall,PhD (Other)
Responsible Party: Sponsor-Investigator, Edward Hall,PhD, Sponsor-Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14-0469-F6A
Record Dates: First submitted 2015-02-03; First posted 2015-07-14 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Cyclosporine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cyclosporine A (Experimental): Participants assigned to this group will receive 2.5mg/kg load then 5mg/kg qd continuous infusion x 3 days (72hours)
  Interventions: Drug: Cyclosporine A
- Placebo (Active Comparator): Participants assigned to this group will receive 2.5mg/kg load then 5mg/kg qd continuous infusion x 3 days (72hours)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Cyclosporine A — Participants will receive 2.5mg/kg load then 5mg/kg qd continuous infusion x 3 days (72hours)
  Arms: Cyclosporine A
Other: Placebo — Participants will receive 2.5mg/kg load then 5mg/kg qd continuous infusion x 3 days (72hours)
  Arms: Placebo

SUMMARY:
This is a prospective, randomized, placebo-controlled study about Cyclosporine A (CSP) and traumatic brain injury (TBI). Cyclosporine A is a drug already marketed and available for other diseases, but is not approved by the Food and Drug Administration for treatment of traumatic brain injury. The effect of Cyclosporine A on chemicals produced following brain injury is being determined using doses no larger than those used for patients having organ transplant. It is also being given for a much shorter time period (3 days). It is not know if side effects seen in patients taking cyclosporine A will occur when it is given for only 3 days. It is not known if patients with brain injury that are treated with cyclosporine A will have side effects like those seen in organ transplant patients.

DETAILED DESCRIPTION:
The purpose of this research study is to measure the chemicals produced by the brain after it is injured and also if Cyclosporine A treatment changes these chemicals. By doing this study, the investigators hope to learn if cyclosporine A therapy helps patients with this injury.

The research procedures will happen at the University of Kentucky (UK) Chandler Medical Center. The study will last for the first 7 days while the participant is admitted to UK Medical Center, or until they are released. Participants will not be asked to stay longer in the hospital for this research study.

Participants in this study will receive all therapies currently available for treatment of severe brain injury. Each participant will be assigned randomly (by chance) to either placebo (a substance without active drug) or cyclosporine A treatment. Neither the participant nor any of the study personnel will know what study treatment has been assigned to the participant.

If assigned to the cyclosporine A treatment group (study drug) participants will be continuously administered the study drug through a tube placed into the vein. A placebo will be given to participants assigned to the placebo group.

Blood and cerebrospinal fluid will be collected at the following time points (12, 24, 36, 48, 60 and 72 hours) for research purposes. These tests will help us understand the participant's ability to make red and white blood cells to fight infection, how well their kidneys function, how well their liver functions, and triglyceride/cholesterol levels.

Cerebrospinal fluid will only be collected from participants who have a drain catheter placed as part of their routine care.

Daily blood collections will occur so the investigators can measure how much of the study drug is present, to assess the body chemicals from the brain and also for safety. Blood samples will be collected by using an already placed line through a vein or artery, or by puncturing the skin with a needle. The chemicals will be measured daily in the urine and also any fluid draining from the line placed into the head for medical management for up to 7 days.

Any unexpected events (side effects) possibly caused by cyclosporine A will be noted and medically managed by the physician. The investigators will be notified when there is need for intervention.

After up to three days of continuous dosing, the study drug will be stopped, but the participant will continue to be carefully monitored for up to 7 days, or until they are released.

Participants will receive the usual treatment for severe traumatic brain injury in addition to receiving the cyclosporine A treatment or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Participant is between the ages of 18 and 65
* Participant speaks and understands English
* CT Scan evidence of severe TBI
* Post resuscitation GSC 4-8 with at least one reactive pupil
* motor score of greater than 5
* Study medication will be administered within 8 hours injury

Exclusion Criteria:

* Participant received high dose systemic corticosteroids, such as Methylprednisolone >15 mg/kg or equivalent,
* Participant has a known allergy to cyclosporine A,
* Participant is pregnant,
* Participant is less than 18 years of age or greater than 65 years of
* Participant has a history of kidney problems, history of stroke or spinal cord injury,
* Participant has a history of cardiovascular disease, or use of immunosuppressive therapy in the last three months,
* Participant has a history of malignant tumors unless they have been in remission at least five years.
* Participant has an active infection
* Participant has taken part in another investigational trial within the last 30 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2017-08-07 (Actual); Study Completion 2017-08-07 (Actual)

PRIMARY OUTCOMES:
Serum lipid peroxidation products: isoprostanes and neuroprostaneses measured by gas-chromatography with mass spectometry | first 7 days after TBI
  Serum lipid peroxidation products will be measured by gas-chromatography with mass spectometry
Cerebrospinal fluid (CSF) calpain-mediated cytoskeletal breakdown products measured by western blotting | first 7 days after TBI
  cytoskeletal breakdown products will be measured by western blotting

SECONDARY OUTCOMES:
ICP Therapy Intensity Level (TIL) Summary | first 7 days after TBI
  The intensity of the use of therapeutic maneuvers to maintain intracranial pressure levels below 20 mm Hg

CONTACTS AND LOCATIONS:
Overall Officials: Edward Hall, PhD, Principal Investigator — Sponsor-Investigator
Locations (1):
- University of Kentucky Medical Center, Lexington, Kentucky, United States

REFERENCES:
- [Background] Hatton J, Rosbolt B, Empey P, Kryscio R, Young B. Dosing and safety of cyclosporine in patients with severe brain injury. J Neurosurg. 2008 Oct;109(4):699-707. doi: 10.3171/JNS/2008/109/10/0699. PMID 18826358